CLINICAL TRIAL: NCT02481960
Title: A Phase I/II Multi Centre Single Arm, Open Label Study of Intraparenchymal Therapy With Irinotecan Hydrochloride Drug-eluting Beads (CM-BC2) as a Adjunct Therapy to Best Standard of Care in Patients With Recurrent, Surgically Resectable High Grade Glioma
Brief Title: Study of Intraparenchymal Therapy With Irinotecan Drug Eluting Beads as Adjunct to Recurrent Surgically Resectable High Grade Glioma
Acronym: IDEB-glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The decision to terminate the trial was based on the slow rate of recruitment across the programme of studies]
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA1018
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Intraparenchymal administration of CM-BC2 irinotecan drug-eluting bead in recurrent high grade glioma.
  Interventions: Procedure: CM-BC2 Irinotecan drug-eluting bead

INTERVENTIONS:
Procedure: CM-BC2 Irinotecan drug-eluting bead
  Other Names: IDEB

SUMMARY:
A study to demonstrate safety, and feasibility for intraparenchymal injection of irinotecan hydrochloride drug-eluting beads in the treatment of recurrent high grade glioma (HGG).

DETAILED DESCRIPTION:
CM-BC2, irinotecan hydrochloride drug-eluting bead, is an investigational product being developed for direct injection in the tumor resection margin, in patients with recurrent high grade glioma (HGG), in order to prevent or delay tumor progression or recurrence.

Patients will be enrolled and receive CM-BC2 following surgical resection of the recurrent high grade glioma and will attend specified study visits until 6 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of Glioblastoma Multiforme (GBM) (World Health Organization grade III or IV)
2. Patient will be considered a good candidate for resection and will have estimated life expectancy of at least 12 weeks as estimated by the Principal Investigator or designee. The decision to opt for resection of the recurrence must be independent of study selection.
3. Tumour characteristics:

   * Single unilateral and supratentorial lesion
   * On clinician's assessment, must be operable under normal considerations of risk vs. benefit for condition and prognosis
4. Patient will have received conventional treatment at the time of initial diagnosis, including surgery (biopsy or de-bulking), and/or radiotherapy, and/or chemotherapy
5. Male or female; no racial exclusions; at least 18 years of age
6. Pregnancy must be excluded in female patients by beta- HCG (Human Chorionic Gonadotropin); all patients agree to use adequate contraception for study duration, not become pregnant or father children during the study
7. Karnofsky Performance Status of at least 50
8. Patients must be able to understand consent and study instructions as well as follow prescribed instructions
9. Patient must have signed written informed consent prior to study participation

Exclusion Criteria:

1. Patient must not be enrolled in any other clinical trial for 30 days before or after participation in this trial
2. History of allergic reactions attributed to compounds of similar chemical make-up or composition to CM-BC2, alginate or irinotecan; or has any other contraindications to irinotecan therapy
3. Open communication between the ventricle CSF (cerebrospinal fluid) and tumour resection cavity/site must be avoided. In the case of opening ventricles during surgery, the surgeon must decide whether effective closure is possible by obstructing the gap with Gelfoam/other appropriate materials
4. Tumor surgery, other than stereotactic biopsy of the high grade glioma, or other neurosurgery within 30 days prior to study entry
5. Irinotecan chemotherapy within 30 days prior to study treatment
6. Radiotherapy or stereotactic (gamma knife) radiosurgery within 90 days prior to study entry
7. Loco-regional (intra-cranial) therapy for the treatment of high grade glioma, including administration of biodegradable polymer wafers containing Carmustine and/or brachytherapy, in the 6 months prior to study entry
8. Significant liver function impairment: aminotransferase (AST) or alanine transaminase (ALT) greater than 2.5 x the upper limit of normal (ULN), or total bilirubin greater than 2 x ULN
9. Significant renal impairment: creatinine greater than 2.0 mg/dL
10. Coagulopathy Prothrombin time (PT) or partial thromboplastin time (APTT) of less than 1.5 x control, and/or platelet count of less than 100 x 10⁹/L
11. Hb less than 8 g/dL and/or neutrophil count (ANC - Absolute Neutrophil Count) of less than 1 x 10⁹/L
12. Any condition that, in the investigator's opinion, makes it in the patient's best interest not to participate in the study
13. Pre-existing cerebral oedema that, in the surgeon's opinion, poses unacceptable risk of post-operative oedema. This decision may be at time of surgery.
14. Presence of concurrent malignancy, except for adequately controlled limited basal cell carcinoma of the skin or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Safety measured by incidence of adverse events as assessed by CTCAE v4 | 6 months
  safety as measured by adverse events including changes in physical exams, neurological function

SECONDARY OUTCOMES:
Progression-free survival | Progression-free survival at 6 months
  progression as assessed by MRI and date of death
Serum levels of irinotecan | 6 months
  serum levels of drug (irinotecan)
Serum levels of SN-38, irinotecan metabolite | 6 months
  serum levels of drug metabolite (SN-38)

CONTACTS AND LOCATIONS:
Locations (2):
- Centre Hopsitalier Universitaire d'Angers, Angers, France
- Prof. Erol Sandalcioglu, Hanover, Germany